CLINICAL TRIAL: NCT00000427
Title: Anabolic Actions of Parathyroid Hormone in Osteoporotic Men
Brief Title: Effects of Parathyroid Hormone in Men With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Joel S. Finkelstein, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50AR044855 (NIH); P50AR044855 (NIH); NIAMS-015
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis
Keywords: Parathyroid Hormone (PTH); Alendronate; Bone metabolism; Bone mineral density (BMD); Bone loss; Postmenopausal osteoporosis; Osteoporosis in men
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — Parathyroid Hormone; Alendronate

INTERVENTIONS:
Drug: Parathyroid hormone
Drug: Alendronate

SUMMARY:
Alendronate is a drug that blocks or reduces bone loss, while parathyroid hormone (PTH) stimulates the formation of new bone. The purpose of this study is to compare the bone-building effects of PTH alone, alendronate alone, and both PTH and alendronate in men with osteoporosis over a two-and-a-half year period.

DETAILED DESCRIPTION:
Osteoporosis causes bones to weaken and break more easily. Alendronate is used to treat or prevent osteoporosis. PTH is a protein hormone that increases the calcium and phosphorus release from bone, leading to formation of new bone. This study will examine the changes in bone density measured at multiple places in the skeleton and changes in chemicals in the body that indicate bone breakdown and bone formation. The study will indicate whether some breakdown of bone is required for PTH to have an overall bone-building effect in men.

Participants will be randomly assigned to receive PTH alone by daily injection under the skin, alendronate alone taken by mouth, or both PTH and alendronate. The study will last 2.5 years. All participants will receive some form of treatment for osteoporosis. Blood, urine, and bone density tests will be performed at 6-month intervals. During the first 6 months, participants will come in for additional study visits.

Participants who complete the initial 2.5 years of their assigned treatment will be eligible for a 12 month extension to monitor bone density and bone turnover after PTH is stopped. Participants who were receiving alendronate will continue taking alendronate. The goal of this extension is to determine what happens to bone density and turnover after PTH is stopped and whether alendronate is needed to prevent loss of PTH-induced bone gain.

Participants who complete the 12 month extension while on their assigned treatment will be eligible for a second 12 month extension in which all participants receive PTH therapy. Participants who have been receiving alendronate continue taking alendronate. The goal of the second extension is to determine if responsiveness to PTH is enhanced by a 12 month suspension of PTH treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bone density of the spine or femoral neck two standard deviations below the mean of young adult men
* Normal renal and liver function tests, normal serum testosterone level, normal vitamin D and PTH levels

Exclusion Criteria:

* Significant cardiac, renal, hepatic, or malignant disease.
* Disorders (e.g., Paget's disease, hyperthyroidism, hyperparathyroidism) or drugs (e.g., steroids, anticonvulsants, lithium, bisphosphonates, calcitonin, fluoride) known to affect bone metabolism
* Active peptic ulcer disease or severe reflux

Ages: 46 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81
Dates: Start 1999-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel S. Finkelstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Finkelstein JS, Klibanski A, Schaefer EH, Hornstein MD, Schiff I, Neer RM. Parathyroid hormone for the prevention of bone loss induced by estrogen deficiency. N Engl J Med. 1994 Dec 15;331(24):1618-23. doi: 10.1056/NEJM199412153312404. PMID 7969342
- [Background] Finkelstein JS, Hayes A, Hunzelman JL, Wyland JJ, Lee H, Neer RM. The effects of parathyroid hormone, alendronate, or both in men with osteoporosis. N Engl J Med. 2003 Sep 25;349(13):1216-26. doi: 10.1056/NEJMoa035725. Epub 2003 Sep 20. PMID 14500805
- [Result] Finkelstein JS, Leder BZ, Burnett SM, Wyland JJ, Lee H, de la Paz AV, Gibson K, Neer RM. Effects of teriparatide, alendronate, or both on bone turnover in osteoporotic men. J Clin Endocrinol Metab. 2006 Aug;91(8):2882-7. doi: 10.1210/jc.2006-0190. Epub 2006 May 9. PMID 16684825